CLINICAL TRIAL: NCT00019812
Title: Study of Trastuzumab (Herceptin) and Paclitaxel in Patients With HER2-Overexpressing Metastatic Breast Cancer
Brief Title: Monoclonal Antibody Plus Chemotherapy in Treating Patients With Metastatic Breast Cancer That Overexpresses HER2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 990121; 99-C-0121; NCI-T98-0087; CDR0000067227; NCT00001819 (obsolete NCT alias)
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2012-03-23 (Estimated); Status verified 2003-04

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; male breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Trastuzumab; Paclitaxel

INTERVENTIONS:
Biological: trastuzumab
Drug: paclitaxel

SUMMARY:
RATIONALE: Monoclonal antibodies such as trastuzumab can locate tumor cells and deliver tumor-killing substances to them without harming normal cells. Drugs used in chemotherapy use different ways to make tumor cells stop dividing so they stop growing or die. Combining monoclonal antibody therapy with chemotherapy may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of trastuzumab plus paclitaxel in treating patients who have metastatic breast cancer that overexpresses HER2.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the pharmacokinetics and pharmacodynamics of trastuzumab (Herceptin) and paclitaxel in patients with HER2-overexpressing metastatic breast cancer.
* Provide access to trastuzumab and paclitaxel for these patients.

OUTLINE: Patients receive trastuzumab (Herceptin) IV over 30-90 minutes and paclitaxel IV over 1 hour weekly. Patients receive trastuzumab alone during course 1 and then in combination with paclitaxel during subsequent courses. Courses repeat every 4 weeks until patients achieve a sustained complete response of 8 weeks or disease progression occurs.

PROJECTED ACCRUAL: A total of 55 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed metastatic breast cancer with HER2 overexpression
* Radiographically or physically measurable disease that can be biopsied safely under local anesthesia
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Male or female

Menopausal status:

* Not specified

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Neutrophil count at least 1,000/mm^3
* Platelet count at least 75,000/mm^3

Hepatic:

* Bilirubin no greater than 3 times upper limit of normal (ULN)
* AST and ALT no greater than 5 times ULN

Renal:

* Not specified

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior trastuzumab

Chemotherapy:

* Not specified

Endocrine therapy:

* At least 2 weeks since prior hormonal therapy
* No concurrent hormone receptor therapy (e.g., tamoxifen or armidex)

Radiotherapy:

* Localized palliative external beam radiotherapy allowed

Surgery:

* Not specified

Other:

* Concurrent bisphosphonates allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 1999-08; Study Completion 2004-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan E. Bates, MD, Principal Investigator — National Cancer Institute (NCI)
Locations (3):
- United States (3):
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - Mary Babb Randolph Center, Morgantown, West Virginia